CLINICAL TRIAL: NCT04329676
Title: A Prospective, Multi-center, Post-market Clinical Follow-up Study of the directSTIM Deep Brain Stimulation (DBS) System
Brief Title: directSTIM Deep Brain Stimulation System Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aleva Neurotherapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-12011
Record Dates: First submitted 2020-03-13; First posted 2020-04-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; DBS; PD
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Patients will undergo bilateral implant of directSTIM system in the STN.
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Patients with PD who are eligible to bilateral STN DBS surgery and chose to get directSTIM System implanted will be followed over a 6-month period to evaluate changes in their condition.

SUMMARY:
The purpose of this study is to obtain clinical outcome data on safety and effectiveness of the directSTIM DBS system when used on-label, according to the instructions for use.

All participants will undergo bilateral implant in the subthalamic nucleus (STN) and data collected in common practice will be recorded during six months post-implant and analyzed.

DETAILED DESCRIPTION:
directSTIM DBS Therapy for Movement Disorders is indicated for patients with disabling tremor or symptoms of Parkinson's disease.

Subjects selected to participate in the study will be Parkinson's Disease (PD) patients who are eligible for bilateral DBS for STN therapy and meet the inclusion criteria and none of the exclusion criteria.

Primary safety and effectiveness endpoints data will be collected through 6 months of follow-up. The values used for comparison are derived from a review of literature spanning from 2001 to 2019.

After completing the 6 month follow-up, subject will exit the study, and continue to be followed by their physician per usual care.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of idiopathic Parkinson's Disease for 4 years or more according to the United Kingdom Parkinson's disease Brain Bank criteria, with disabling motor complications despite optimal medical treatment.
* Patient is eligible for bilateral DBS for STN therapy according to center's routine criteria and according to the directSTIM DBS system Indications for Use statement.
* Patient who is willing to provide a written informed consent.
* Patient complies with the study follow-up, in particular the follow-up visits, and other study requirements.

Exclusion Criteria:

* Patient is not eligible for DBS per center criteria.
* Patient has a cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to complete study assessments, such as:

  * Active major psychiatric disorder.
  * Dementia (MoCa Dementia Rating Scale score <26 or otherwise not capable of discernment).
  * Presence of an electrical or electromagnetic implant (e.g. cochlear implant, pacemaker).
  * Previous surgery for the treatment of Parkinson's disease.
  * Previous brain ablation procedure.
  * Epilepsy.
  * Coagulopathies.
  * Abuse of drugs or alcohol.
* Patient is participating in another clinical study that would confound data analysis.
* Patient is pregnant or nursing. As for other DBS systems, the effects of the device on an unborn child are not established.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in UPDRS III score without medication | 6 months compared to baseline
  Part 3 of the Unified Parkinson's Disease Rating Scale (UPDRS III), is a series of questions evaluated by the clinician in presence of the patient, focusing on motor symptoms of PD.
  Score is expressed on a scale of 0 to 108. This score is evaluated at baseline and 6 months post-implant without any anti-Parkinson medication taken.
  A decrease at 6 months compared to baseline indicates an improvement. The average difference of scores between the two time points is calculated for the whole study subject population.
  This value is to be compared to the results of a meta-analysis performed on data extracted during a literature search.
Materiovigilance | 6 months
  Summary statistics on the occurrence of the following categories of adverse events (AEs):
  * Device-related AEs
  * Procedure-related AEs
  * Stimulation-related AEs

SECONDARY OUTCOMES:
Therapeutic Window (TW) | 3 months
  The therapeutic window is the difference of electrical current values between the stimulation settings that provide maximum alleviation of motor symptoms and the settings for which the first stimulation-induced side effect appears (e.g., eye deviation, muscle contraction, speech impairment).
  The wider this window, the more flexibility is offered to the patient for stimulation without causing side-effects.
UPDRS | 6 months
  Other parts (I, II and IV) of the Unified Parkinson's Disease Scale are evaluated at baseline and 6 months post-implant.
  Part I is a series of 4 questions assessing Mentation, Behavior and Mood. Patient's score is expressed on a scale of 0 to 16.
  Part II is a series of 13 questions assessing Quality of Life in daily activities. Patient's score is expressed on a scale of 0 to 52.
  Part IV is a series of 10 questions assessing Complications of Therapy. Patient's score is expressed on a scale of 0 to 23.
  A decrease at 6 months compared to baseline indicates an improvement.

OTHER OUTCOMES:
Change in PDQ-39 score | 6 months
  Parkinson's Disease Questionnaire-39, a patient-filled questionnaire focusing on quality of life, is completed by study subjects at baseline and 6 months post-implant.
  Score is expressed on a scale of 0 to 100. A decrease at 6 months compared to baseline indicates an improvement.
  The average difference of scores between the two time points is calculated for the whole study subject population.
Change in dopaminergic medication | 6 months
  The Levodopa equivalent daily dose (LEDD) is expressed as Levodopa equivalent mg/day and measured through the whole study duration.
  Evolution of this value is followed and the difference between baseline and 6 months post-implant timepoints is to be compared to the results of a meta-analysis performed on data extracted during a literature search.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Dransart, Study Director — Aleva Neurotherapeutics SA
Locations (6):
- Germany (6):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein (Kiel), Kiel
  - Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: No
Principal Investigator
  The principal investigator will publish and/or present the data generated from the clinical investigation, following the conditions specified in the Clinical Site Agreement.
  Sponsor
  Sponsor will use this data for internal monitoring of product safety and performance for regulatory purposes, by performing regular updates of the safety profile and the planned interim analyses.